CLINICAL TRIAL: NCT04311099
Title: Laparoscopic vs Ultrasound-Guided Transversus Abdominis Plane Block in Minimally Invasive Colon Surgery: A Randomized Controlled Multicentre Clinical Trial
Brief Title: Optimal Peripheral Nerve Block After Minimally Invasive Colon Surgery
Acronym: OPMICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claus Anders Bertelsen, PhD, MD (Other)
Responsible Party: Sponsor-Investigator, Claus Anders Bertelsen, PhD, MD, Associate professor, consultant surgeon, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPMICS-1
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Pain, Abdominal; Analgesia; Surgery; Colon Cancer; Injection Site
MeSH Terms: conditions — Pain, Postoperative; Abdominal Pain; Agnosia; Colonic Neoplasms | interventions — Bulk Drugs; Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ultrasound-guided TAP (Experimental): Ultrasound-guided TAP with 20 ml ropivacaine 2 mg/ml solution bilaterally and laparoscopic assisted injection of 20 ml saline (placebo) bilaterally at the beginning of surgery
  Interventions: Drug: Active drug; Drug: Placebo; Procedure: Injection of Ropivacaine - Ultrasound-guided transverse abdominal plane block; Procedure: Injection of placebo - Laparoscopic assisted transverse abdominal plane block
- Laparoscopic assisted TAP (Experimental): Laparoscopic assisted TAP with 20 ml ropivacaine 2 mg/ml solution bilaterally and ultrasound-guided injection of 20 ml saline (placebo) bilaterally at the beginning of surgery
  Interventions: Drug: Active drug; Drug: Placebo; Procedure: Injection of Ropivacaine - Laparoscopic assisted transverse abdominal plane block; Procedure: Injection of placebo - Ultrasound-guided transverse abdominal plane block
- Placebo (Placebo Comparator): Laparoscopic assisted injection of 20 ml saline (placebo) bilaterally and ultrasound-guided injection of 20 ml saline (placebo) bilaterally at the beginning of surgery
  Interventions: Drug: Placebo; Procedure: Injection of placebo - Ultrasound-guided transverse abdominal plane block; Procedure: Injection of placebo - Laparoscopic assisted transverse abdominal plane block

INTERVENTIONS:
Drug: Active drug — Injection of Ropivacaine
  Other Names: Ropivacaine
  Arms: Laparoscopic assisted TAP; Ultrasound-guided TAP
Drug: Placebo — Injection of Saline solution
  Other Names: Saline solution
Procedure: Injection of Ropivacaine - Ultrasound-guided transverse abdominal plane block — Lateral ultrasound-guided transverse abdominal plane block 40 ml ropivacaine 2 mg / ml
  Arms: Ultrasound-guided TAP
Procedure: Injection of Ropivacaine - Laparoscopic assisted transverse abdominal plane block — Laparoscopic assisted subcostal transverse abdominal plane block 40 ml ropivacaine 2 mg / ml
  Arms: Laparoscopic assisted TAP
Procedure: Injection of placebo - Ultrasound-guided transverse abdominal plane block — Lateral ultrasound-guided transverse abdominal plane block with saline solution
  Arms: Laparoscopic assisted TAP; Placebo
Procedure: Injection of placebo - Laparoscopic assisted transverse abdominal plane block — Laparoscopic assisted subcostal transverse abdominal plane block with saline solution
  Arms: Placebo; Ultrasound-guided TAP

SUMMARY:
The purpose of the trial is to identify the "most simple non-inferior of three different methods", placebo, laparoscopic assisted transverse abdominal plane block (L-TAP) and ultrasound guided TAP block (US-TAP), using postoperative opioid consumption as a measure of efficacy in patients undergoing elective minimally invasive colon surgery in an ERAS setting. Postoperative pain scores and length of stay (LOS) will also be measured. The simplicity of the three methods is ranked as: 1) placebo, 2) L-TAP and 3) US-TAP.

DETAILED DESCRIPTION:
Introducing laparoscopy in colorectal surgery and optimizing the postoperative care using the standardized protocols of enhanced recovery after surgery (ERAS) have significantly improved patient outcomes and LOS. Better pain management has the potential to further improve these outcomes. Since the introduction of ultrasound-guided abdominal wall blocks, much research has been done in that field, but no consensus has been reached concerning the optimal block technique; where to and when to inject the block, or which drug to use. Newly published randomized controlled trials show interesting results regarding the L-TAP which has several advantages to the US-TAP, including the ease of performance, less dependency on specialized skills or equipment and avoidance of intraperitoneal infiltration. but these results need to be solidified with multicentre trials. Besides optimizing postoperative pain management, better block techniques could potentially decrease LOS in patients after minimally invasive colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to receive curative elective minimally invasive colon surgery for colon cancer or adenoma without a planned ostomy. Colon cancer or adenoma is defined by a distance of more than 15 cm from the anal verge to the distal limitation of the tumour or adenoma as measured by rigid sigmoidoscope. The following procedural codes are included:
* Laparoscopic ileocecal resection
* Laparoscopic right hemicolectomy
* Other laparoscopic resection of both small and large bowel
* Laparoscopic resection of transverse colon
* Laparoscopic left hemicolectomy
* Laparoscopic resection of sigmoid colon
* Other laparoscopic colon resection
* Having given informed written consent.

Exclusion Criteria:

* Known allergy to local analgesics
* Known liver failure Class C according to the Child-Pugh Score
* Body weight of less than 40 kg
* History of being a chronic pain patient (weekly intake WHO step II or step III or adjuvant step I analgesic)
* Presence of concomitant painful conditions other than low back pain that could confound the subject's trial assessments or self-evaluation of the index pain, e.g., syndromes with widespread pain such as fibromyalgia
* Predictably non-compliant due to language barrier or psychiatric disease
* Patients rescheduled for open surgery, before the intervention has been administered
* Patients where the indication for surgery changes before the intervention has been administered
* Patients with known inflammatory bowel disease
* Patients who have previously undergone open major abdominal surgery defined by prior intraabdominal surgery with a midline or upper abdominal incision of more than 8 cm
* Incisional hernia
* Patients with a history of abdominal wall surgery including resection of the external oblique muscles, the internal oblique muscles, the transversus abdominis muscles, the rectus abdominis muscles or their fascial components
* Pregnancy (patients are screened using urine human chorionic gonadotropin upon admission if female and not postmenopausal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Total morphine dose equivalents administered. | The first 24 hours from the end of anesthesia.
  Intravenously in milligrams.

SECONDARY OUTCOMES:
Total morphine dose equivalents administered in the operation theater. | Up to 12 hours.
  Intravenously in milligrams.
Total morphine dose equivalents administered in the post anesthesia care unit. | The first 24 hours from the end of anesthesia.
  Intravenously in milligrams.
Postoperative pain at rest - 8:00-10:00 AM (ante meridiem) Postoperative Day 1. | Postoperative Day 1.
  11-point Numeric Rating Scale. 0-10 (higher score - worse outcome).
Postoperative pain when coughing - 8:00-10:00 AM Postoperative Day 1 | Postoperative Day 1.
  11-point Numeric Rating Scale. 0-10 (higher score means worse outcome)
Postoperative length of stay. | Up to 30 days.
  Days - Measured from the end of anesthesia.
Incidence of Postoperative Nausea and Vomiting - 8:00-10:00 AM Postoperative Day 1. | Postoperative Day 1.
  4-point Numeric Rating Scale. 0-3 (higher score means worse outcome).
Total dose of antiemetic medication administered. | In the first 24 hours from the end of anesthesia.
  Intravenously in milligrams.
Total dose of antiemetic medication administered in the operating theater. | Up to 12 hours.
  Intravenously in milligrams.
Time spent in the post anesthesia care unit. | Up to 30 hours.
  From the end of anesthesia to discharge to ward. Measured in hours and minutes.
Postoperative mobilisation. | Postoperative Day 1.
  4-point Verbal Rating Scale. 1-4 (higher score means worse outcome).
Quality of Recovery 15. | Postoperative Day 1.
  The Quality of Recovery 15 is a 15-item questionnaire that measures the patient's quality of recovery. Each item is answered on an 11-point Numerical Rating Scale. The score ranges from 0 to 150 with a higher score indicating a better quality of recovery. It measures in the domains of pain, physical comfort, physical independence, psychological support, and emotional state.
Postoperative complications. | Postoperative Day 30.
  According to the Clavien-Dindo classification of surgical complications.
Need for rescue TAP-block or epidural analgesia. | Postoperative Day 30.
  Epidural or TAP-block administered post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, Study Chair — Copenhagen University Hospital - North Zealand
Locations (5):
- Denmark (5):
  - Sydvestjysk Sygehus, Esbjerg
  - Regionshospitalet Herning, Herning
  - Copenhagen University Hospital - North Zealand, Hillerød
  - Copenhagen University Hospital - Hvidovre, Hvidovre
  - Regionshospitalet Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Yes
After de-identification, individual participant data will be made available to investigators who provide a methodologically sound proposal for meta-analyses. Proposals should be directed to Claus A Bertelsen (cabertelsen@gmail.com). A Data Processing Agreement according to the EU General Data Protection Regulation has to be signed before data sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 15 years after publication
Access Criteria: A methodologically sound proposal for meta-analyses

REFERENCES:
- [Background] Lund H, Spanager L, Winther ACR, Gierloff M, Sunekaer K, Kleif J, Bertelsen CA. Recurrence and complications after laparoscopic inguinal hernia repair using a self-adherent mesh: a patient-reported follow-up study. Surg Endosc. 2025 Apr;39(4):2464-2470. doi: 10.1007/s00464-025-11614-7. Epub 2025 Feb 24. PMID 39994048
- [Background] Salmonsen CB, Lange KHW, Kleif J, Kroijer R, Bruun L, Mikalonis M, Dalsgaard P, Hesseldal KB, Olsson JEP, Bertelsen CA; OPMICS Study Group. Transversus abdominis plane block in minimally invasive colon surgery: a multicenter three-arm randomized controlled superiority and non-inferiority clinical trial. Reg Anesth Pain Med. 2025 Jan 23:rapm-2024-105712. doi: 10.1136/rapm-2024-105712. Online ahead of print. PMID 39542642
- [Background] Helander EM, Webb MP, Bias M, Whang EE, Kaye AD, Urman RD. A Comparison of Multimodal Analgesic Approaches in Institutional Enhanced Recovery After Surgery Protocols for Colorectal Surgery: Pharmacological Agents. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):903-908. doi: 10.1089/lap.2017.0338. Epub 2017 Jul 25. PMID 28742427
- [Background] Grant MC, Yang D, Wu CL, Makary MA, Wick EC. Impact of Enhanced Recovery After Surgery and Fast Track Surgery Pathways on Healthcare-associated Infections: Results From a Systematic Review and Meta-analysis. Ann Surg. 2017 Jan;265(1):68-79. doi: 10.1097/SLA.0000000000001703. PMID 28009729
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Neal JM, Brull R, Chan VW, Grant SA, Horn JL, Liu SS, McCartney CJ, Narouze SN, Perlas A, Salinas FV, Sites BD, Tsui BC. The ASRA evidence-based medicine assessment of ultrasound-guided regional anesthesia and pain medicine: Executive summary. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S1-9. doi: 10.1097/AAP.0b013e3181d22fe0. PMID 20216019
- [Background] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Background] Keller DS, Madhoun N, Ponte-Moreno OI, Ibarra S, Haas EM. Transversus abdominis plane blocks: pilot of feasibility and the learning curve. J Surg Res. 2016 Jul;204(1):101-8. doi: 10.1016/j.jss.2016.04.012. Epub 2016 Apr 27. PMID 27451874
- [Background] Keller DS, Ermlich BO, Schiltz N, Champagne BJ, Reynolds HL Jr, Stein SL, Delaney CP. The effect of transversus abdominis plane blocks on postoperative pain in laparoscopic colorectal surgery: a prospective, randomized, double-blind trial. Dis Colon Rectum. 2014 Nov;57(11):1290-7. doi: 10.1097/DCR.0000000000000211. PMID 25285696
- [Background] Favuzza J, Brady K, Delaney CP. Transversus abdominis plane blocks and enhanced recovery pathways: making the 23-h hospital stay a realistic goal after laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2481-6. doi: 10.1007/s00464-012-2761-y. Epub 2013 Jan 26. PMID 23355160
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Chetwood A, Agrawal S, Hrouda D, Doyle P. Laparoscopic assisted transversus abdominis plane block: a novel insertion technique during laparoscopic nephrectomy. Anaesthesia. 2011 Apr;66(4):317-8. doi: 10.1111/j.1365-2044.2011.06664.x. No abstract available. PMID 21401554
- [Background] Elamin G, Waters PS, Hamid H, O'Keeffe HM, Waldron RM, Duggan M, Khan W, Barry MK, Khan IZ. Efficacy of a Laparoscopically Delivered Transversus Abdominis Plane Block Technique during Elective Laparoscopic Cholecystectomy: A Prospective, Double-Blind Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):335-44. doi: 10.1016/j.jamcollsurg.2015.03.030. Epub 2015 Mar 27. PMID 25899736
- [Background] Park SY, Park JS, Choi GS, Kim HJ, Moon S, Yeo J. Comparison of Analgesic Efficacy of Laparoscope-Assisted and Ultrasound-Guided Transversus Abdominis Plane Block after Laparoscopic Colorectal Operation: A Randomized, Single-Blind, Non-Inferiority Trial. J Am Coll Surg. 2017 Sep;225(3):403-410. doi: 10.1016/j.jamcollsurg.2017.05.017. Epub 2017 Jun 10. PMID 28610880
- [Background] Zaghiyan KN, Mendelson BJ, Eng MR, Ovsepyan G, Mirocha JM, Fleshner P. Randomized Clinical Trial Comparing Laparoscopic Versus Ultrasound-Guided Transversus Abdominis Plane Block in Minimally Invasive Colorectal Surgery. Dis Colon Rectum. 2019 Feb;62(2):203-210. doi: 10.1097/DCR.0000000000001292. PMID 30540660
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Dickerson DM, Apfelbaum JL. Local anesthetic systemic toxicity. Aesthet Surg J. 2014 Sep;34(7):1111-9. doi: 10.1177/1090820X14543102. Epub 2014 Jul 15. PMID 25028740
- [Background] Naidu RK, Richebe P. Probable local anesthetic systemic toxicity in a postpartum patient with acute Fatty liver of pregnancy after a transversus abdominis plane block. A A Case Rep. 2013 Dec 1;1(5):72-4. doi: 10.1097/ACC.0b013e3182973a2f. PMID 25612087
- [Background] Statzer N, Cummings KC 3rd. Transversus Abdominis Plane Blocks. Adv Anesth. 2018 Dec;36(1):163-180. doi: 10.1016/j.aan.2018.07.007. Epub 2018 Sep 27. No abstract available. PMID 30414636
- [Background] Chin KJ, McDonnell JG, Carvalho B, Sharkey A, Pawa A, Gadsden J. Essentials of Our Current Understanding: Abdominal Wall Blocks. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):133-183. doi: 10.1097/AAP.0000000000000545. PMID 28085788
- [Background] Sullivan MJL, Bishop SR, Pivik J. The pain catastrophizing scale: development and validation. Psychol Assess 1995; 7: 524.
- [Derived] Salmonsen CB, Lange KHW, Kleif J, Bertelsen CA. Optimal peripheral nerve block after minimally invasive colon surgery - a study protocol for a randomised trial. Dan Med J. 2021 Nov 12;68(12):A03210245. PMID 34851250